CLINICAL TRIAL: NCT00345631
Title: ECLIPSE Trial - Ensure's Vascular Closure Device Speeds Hemostasis Trial
Brief Title: Safety and Effectiveness Study of the Ensure Medical Vascular Closure Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Chao-Chin Chen, Vice President, Ensure Medical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM0501
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Arteriosclerosis; Peripheral Arteriosclerosis
Keywords: Closure Device; Angiography; Angioplasty; Hemostasis; Heart Catheterization; Peripheral Angiography; Femoral Closure; Vascular Closure; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Vascular Closure Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual Compression (Active Comparator): Manual compression (MC)
  Interventions: Other: Manual Compression
- Vascular Closure Device (Experimental): Vascular Closure Device (VCD)
  Interventions: Device: Vascular Closure Device

INTERVENTIONS:
Other: Manual Compression — Manual compression
  Arms: Manual Compression
Device: Vascular Closure Device — Investigational vascular closure device
  Other Names: Exoseal
  Arms: Vascular Closure Device

SUMMARY:
The purpose of this study is to determine whether the Ensure Medical Vascular Closure Device is more effective than standard manual compression at sealing the puncture made in the femoral artery following a cardiac or peripheral diagnostic or interventional procedure while maintaining the same level of safety.

DETAILED DESCRIPTION:
Achieving hemostasis at the arterial puncture site after percutaneous cardiac catheterization is a potential cause of bleeding, hematomas, pseudoaneurysms, and various other vascular complications. Hemostasis at the femoral artery access site after diagnostic or interventional procedures is typically achieved using either manual compression or the deployment of a vascular closure device. Manual compression is time consuming for the health-care provider, and painful for the patient. In addition, prolonged periods of immobilization and bed rest may be required. Vascular closure devices have been developed to avoid manual compression, shorten bed rest, and allow earlier ambulation.

The Ensure Medical Vascular Closure device (VCD) is intended for femoral artery puncture site closure in patients who have undergone coronary or peripheral diagnostic or interventional procedure using a standard 6F introducer sheath. The device is comprised of a bio-absorbable plug and a plug delivery system. The plug delivery system is designed to position the bio-absorbable plug to the extravascular surface of the femoral artery access site, facilitating a hemostasis response. The Ensure Medical VCD has been studied in a prior feasibility trial of 149 patients, which demonstrated that: (1) the device could be used to successfully obtain rapid hemostasis and early ambulation in patients undergoing catheterization procedures; and (2) the low incidence and relatively minor nature of the observed closure related complications suggests that the device is safe for its intended purpose.

The ECLIPSE Trial is designed to evaluate the safety and effectiveness of the Ensure Medical VCD in comparison to standard manual compression. Patients will be randomly assigned to have their arterial access site closed using either manual compression or the VCD. The principal comparisons of the two closure techniques will include:

* Time required to obtain hemostasis of the vascular access site
* Time required for the patient to ambulate after their catheterization
* Frequency of occurrence of serious closure-related complications

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a coronary or peripheral diagnostic or interventional procedure
* Able to undergo emergent vascular surgery if a complication requires it
* 6F arterial puncture located in the common femoral artery
* Femoral artery has a lumen diameter of at least 5 mm

Exclusion Criteria:

* Arterial puncture in the femoral artery of both legs
* Prior target artery closure with any vascular closure device, or closure with manual compression within 30 days prior to catheterization
* Patients who bruise or bleed easily or with a history of significant bleeding or platelet disorders
* Acute ST-elevation myocardial infarction within 48 hours prior to catheterization
* Uncontrolled hypertension at time of vessel closure
* Elevated Activated Clotting Time at time of vessel closure
* Ineligible for in-catheterization lab introducer sheath removal
* Concurrent participation in another investigational device or drug trial
* Thrombolytic therapy, bivalirudin, other thrombin-specific anticoagulants, or low molecular weight heparin within 24 hours prior to catheterization
* Preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the vessel access site prior to femoral artery closure
* Prior femoral vascular surgery or vascular graft in region of access site
* Femoral artery is tortuous or requires an introducer sheath longer than 11 cm
* Fluoroscopically visible calcium, atherosclerotic disease, or stent within 1 cm of the puncture site that would interfere with the operation of the experimental device
* Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
* Antegrade vascular puncture
* Body Mass Index over 40 kg/m^2
* Symptomatic leg ischemia in the target limb including severe claudication or weak/absent pulse
* Femoral artery diameter stenosis exceeding 50%
* Pre-existing severe non-cardiac systemic disease or terminal illness
* Planned arterial access at the same access site within 30 days of catheterization
* Extended hospitalization (e.g. Coronary Artery Bypass Graft (CABG) surgery)
* Pre-existing systemic or cutaneous infection
* Prior use of an intra-aortic balloon pump through the arterial access site
* Cardiogenic shock during or immediately following the catheterization
* Patient is unable to ambulate at baseline
* Patient is known or suspected to be pregnant or is lactating
* Patient is unavailable for follow-up
* Any angiographic or clinical evidence that the physician feels would place the patient at increased risk with the use of the experimental device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2007-02; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Chiu Wong, MD, Principal Investigator — New York Presbyterian Hospital
Locations (17):
- United States (17):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - Stanford University, Stanford, California
  - Morton Plant Hosptial, Clearwater, Florida
  - The Care Group, Indianapolis, Indiana
  - Washington University School of Medicine at Barnes-Jewish Hospital, St Louis, Missouri
  - Cooper Health Systems, Camden, New Jersey
  - SJH Cardiology Associates, Liverpool, New York
  - New York Presbyterian Hospital - Cornell Medical College of Cornell University, New York, New York
  - Wake Heart Research, Raleigh, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hahnemann Hospital, Philadelphia, Pennsylvania
  - Moffitt Heart & Vascular Group, Wormleysburg, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Result] Wong SC, Bachinsky W, Cambier P, Stoler R, Aji J, Rogers JH, Hermiller J, Nair R, Hutman H, Wang H; ECLIPSE Trial Investigators. A randomized comparison of a novel bioabsorbable vascular closure device versus manual compression in the achievement of hemostasis after percutaneous femoral procedures: the ECLIPSE (Ensure's Vascular Closure Device Speeds Hemostasis Trial). JACC Cardiovasc Interv. 2009 Aug;2(8):785-93. doi: 10.1016/j.jcin.2009.06.006. PMID 19695549

RESULTS

PARTICIPANT FLOW:
Groups:
- Roll-In: Roll-In patients were device training patients
- Vascular Closure Device: Ensure Medical Vascular Closure Device (VCD) have been developed to avoid manual compression, shorten bed rest, and allow earlier ambulation.
- Manual Compression: Traditionally Hemostasis at the femoral artery access site after diagnostic or interventional procedures is typically achieved using either manual compression (with or without the use of adjunctive mechanical compression devices)
Period: Overall Study
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Started | 87 | 267 | 134
Completed | 83 | 259 | 128
Not Completed | 4 | 8 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 7 | 4
Not completed — Other reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression | Total
Number analyzed (Participants) | 87 | 267 | 134 | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 144 | 83 | 274
  >=65 years | 40 | 123 | 51 | 214
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.61) | 63.3 (11.13) | 61.4 (10.47) | 62.8 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 85 | 51 | 165
  Male | 58 | 182 | 83 | 323
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 8 | 18
  Not Hispanic or Latino | 84 | 260 | 126 | 470
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 10 | 23 | 13 | 46
  White | 77 | 236 | 114 | 427
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 87 | 267 | 134 | 488

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis (TTH)
Description: Time to hemostasis is defined as time (in minutes) from when the introducer sheath was removed to the time that hemostasis was first observed during post-procedure follow up. Hemostasis is defined as no or minimal subcutaneous oozing and the absence of expanding or developing hematoma. Time to hemostasis is one of the two co-primary endpoints.
Time Frame: From when the introducer sheath was removed to the time hemostasis was first observed
Population: Intent to treat population (ITT) with non-missing time to hemostasis data. ITT population consists of all randomized (VCD and MC) patients where a femoral artery closure procedure is attempted post-randomization.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Roll-In: patients were device training patients
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 267 | 131
Minutes | 4.68 (19.37) | 4.38 (11.59) | 20.05 (22.54)
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Null hypothesis: The mean time to hemostasis for the manual compression (MC) arm is less or equal to that for the vascular closure device (VCD) arm. The trial is powered to detect a 5 minute reduction in mean time to hemostasis and a 2 hour reduction in mean time to ambulation for VCD vs. MC with over 90% power and a 5% two-sided (2.5% one-sided) Type I error; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Multiplicity is addressed for the two co-primary effectiveness endpoints via a closed testing procedure where the time to hemostasis will be assessed first and then time to ambulation only if significance is first achieved for time to hemostasis; Mean Difference (Net) = -15.68, 95% CI 2-sided [-19.04 to -12.31]

2. Primary Outcome: Time to Ambulation (TTA)
Description: Time to ambulation is defined as the time from when the introducer sheath was removed to the time that ambulation was achieved. Ambulation is defined as patient standing and walking at least 20 feet without re-bleeding or significant oozing requiring manual compression. Time to ambulation is one of the two co-primary endpoints.
Time Frame: From when the introducer sheath was removed to 30 days post-procedure
Population: Intent to Treat (ITT)Population with non-missing time to ambulation data.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 264 | 129
Hours | 1.98 (2.59) | 2.54 (5.02) | 6.24 (13.34)
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Null hypothesis:The mean time to ambulation for the manual compression (MC) arm is less or equal to that for the vascular closure device (VCD) arm. The trial is powered to detect a 5 minute reduction in mean time to hemostasis and a 2 hour reduction in mean time to ambulation for VCD vs. MC with over 90% power and a 5% two-sided (2.5% one-sided) Type I error; Test type: Superiority or Other; p = 0.0028, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -3.70, 95% CI 2-sided [-5.53 to -1.87]

3. Primary Outcome: Percentage of Patients Who Experience Any Vascular Closure Related Major Adverse Events During the 30 Days Post-procedure
Description: Vascular closure related major adverse events consist of any of the events below: Vascular repair or the need for repair; access site-related bleeding requiring transfusion; access site-related infection requiring intravenous/intramuscular antibiotics and/or extended hospitalization; any new ipsilateral lower extremity ischemia documented by symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram; surgery for access site-related nerve injury; and Permanent (> 30 days) access site-related nerve injury.
Time Frame: From post-procedure to 30 days follow up
Population: Intent to treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 267 | 134
Percentage of participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Based on pre-planned hypotheses, a minimum sample size of 390 randomized patients (260 VCD patients and 130 MC patients) would demonstrate non-inferiority for the primary safety endpoint and superiority for both co-primary effectiveness endpoints in comparing VCD vs. MC; Test type: Non-Inferiority or Equivalence — The sample size is adequate to rule out a 4% or larger disadvantage for VCD vs. MC (null hypothesis: 2.5% MC vs. 6.5% VCD) in the incidence of major complications for VCD vs. MC using a 95% upper confidence bound for the VCD - MC difference with 80% power and a 5% one-sided Type I error; p = 0.0006, unconditional exact test — P-value was calculated using unconditional exact test of non-inferiority for difference of two binomial proportions (VCD vs. MC) with a margin of 4%; Mean Difference (Final Values) = 0, 95% CI 1-sided [upper limit 1.14]

4. Secondary Outcome: Time to Eligibility for Hospital Discharge
Description: Time to Eligibility for Hospital Discharge is measured from the time of sheath removal to the time when the patient is eligible for discharge according to the judgment of the patient's physician.
Time Frame: From introducer sheath removal to hospital discharge, up to 284 hours
Population: Intent to treat population with non-missing time data
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 85 | 257 | 128
Hour | 9.72 (14.15) | 12.57 (13.91) | 16.25 (27.49)
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Null hypothesis: The mean time to eligibility for hospital discharge for the manual compression (MC) arm is equal to that for the vascular closure device (VCD) arm; Test type: Superiority or Other; p = 0.1540, t-test, 2 sided; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-7.84 to 0.45]

5. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge is defined as from the time of sheath removal to the time of hospital discharge
Time Frame: From introducer sheath removal to patient discharge
Population: Intent to Treat population with non-missing time data
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 264 | 133
Hour | 13.64 (18.54) | 16.77 (19.79) | 19.35 (29.23)
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Null hypothesis: The mean time to hospital discharge for the manual compression (MC) arm is equal to that for the vascular closure device (VCD) arm; Test type: Superiority or Other; p = 0.3612, t-test, 2 sided; Mean Difference (Final Values) = -2.57, 95% CI 2-sided [-7.46 to 2.31]

6. Secondary Outcome: Time to Device Deployment, up to 5 Minutes
Description: Time to device deployment is defined as from the time device inserted to the time sheath removed
Time Frame: From device inserted to introducer sheath removal
Population: Intent to Treat population with non-missing time data, excluding MC patients. Patients in the MC arm didn't deploy the device.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 260 | 0
Hour | 0.94 (1.13) | 1.01 (2.12) |

7. Secondary Outcome: Percentage of Patients Who Achieved Device Success Within Five Minutes Post-procedure
Description: Device Success is defined as the successful deployment of the plug, initial hemostasis time less or equal to 5 minutes, and removal of the intact delivery system.
Time Frame: Within 5 minutes post-procedure
Population: Intent to treat population (ITT) excluding the Manual Compression (MC) patients since MC Patients didn't deploy the device.
Measure: Number; unit: Percentage of participants
Groups:
- Manual Compression (Not Applicable for Device Success): Traditionally Hemostasis at the femoral artery access site after diagnostic or interventional procedures is typically achieved using either manual compression (with or without the use of adjunctive mechanical compression devices)
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression (Not Applicable for Device Success)
Number analyzed (Participants) | 87 | 267 | 0
Percentage of participants | 95.4 | 89.1 |

8. Secondary Outcome: Percent of Patients Who Achieved Procedure Success During 30 Days Post-procedure
Description: Procedure success is defined as initial hemostasis achieved by the assigned method Vascular Closure Device (VCD) or Manual compression (MC) with none of the primary safety endpoint's closure related major adverse events (MAE). Procedural success is assessed on day of catheterization procedure and at 30 days post-procedure.
Time Frame: From catheterization procedure to 30 day post-procedure follow up
Population: Intent to Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 267 | 134
Percentage of participants | 95.4 | 91.8 | 91.0
Statistical Analysis 1: Comparison: Vascular Closure Device vs Manual Compression; Null hypothesis: The percentages of patients achieving procedure success between the vascular closure device and manual compression arms are equal; Test type: Superiority or Other; p = 0.85, t-test, 2 sided; Proportion difference = 0.7, 95% CI 2-sided [-4.8 to 7.4]

9. Secondary Outcome: Percentage of Patients Who Experienced Any Other Vascular Closure Related Adverse Events
Description: Other known vascular closure related adverse events include: Rebleeding Following Initial Hemostasis; Access Site Hematoma >= 6cm; Access Site-Related Bleeding Requiring > 30 min for Hemostasis; Transient Access Site-Related Nerve Injury; Retroperitonea Bleeding; Decrease in Pedal Pulse
Time Frame: From end of vessel closure procedure to 30 days post-procedure
Population: Intent to treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Number analyzed (Participants) | 87 | 267 | 134
Percentage of participants | 10.3 | 8.99 | 4.48

ADVERSE EVENTS:
Arm/Group | Roll-In | Vascular Closure Device | Manual Compression
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/267 | 0/134
Other Adverse Events (participants affected / at risk) | 7/87 | 24/267 | 6/134
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-In (N=87) | Vascular Closure Device (N=267) | Manual Compression (N=134)
Rebleeding Following Initial Hemostasis (Blood and lymphatic system disorders) | 3 (3) | 14 (14) | 3 (3)
Access Site Hematoma >= 6cm (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 1 (1)
Access Site-Related Bleeding Requiring > 30 min for Hemostasis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Transient Access Site-Related Nerve Injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal Bleeding (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Eochymosis >= 6cm (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Decrease in Pedal Pulse (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days